CLINICAL TRIAL: NCT03876249
Title: The Consequence of Respiratory Syncytial Virus (RSV) Infection in Young Infants
Brief Title: The Long-term Effect of RSV Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Child Health Research Foundation, Bangladesh (Other)
Collaborators: University of Edinburgh (Other); Aga Khan University (Other); Projahnmo Research Foundation (Other); Asian Institute of Public Health (Other); KEM Hospital Research Centre (Other); Maternal, Neonatal and Child Health Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: CHRF001
Record Dates: First submitted 2019-03-02; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Asthma in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RSV positive group: Children who had RSV infection within the first 60 days of life
  Interventions: Other: exposure to RSV
- RSV negative group: Children without known RSV infection within the first 60 days of life
  Interventions: Other: exposure to RSV

INTERVENTIONS:
Other: exposure to RSV — No intervention will be given, children naturally exposed to RSV in their early life

SUMMARY:
Respiratory Syncytial Virus (RSV) is a leading cause of childhood illness and hospitalization across the world. In addition to acute mortality and morbidity, RSV infection is associated with developing recurrent wheeze in pre-school children and asthma in later life. The overarching aim of the study is to demonstrate the long-term effect of RSV infection on child health in resource-poor settings.

Children previously infected with RSV in their first two months of life and age-matched controls will be followed and epidemiological data will be compared in terms of prevalence of asthma, lung function status, physical growth status, and asthma risk factors. Enrolled children will be routinely assessed for a period of 12 months. During this period, this study will record the health status of the children (respiratory tract illness, wheeze, cough, other illness, and attendance at medical services), physical growth (height, weight and mid-upper arm circumference), family history of atopic diseases (e.g. asthma) and environmental risk exposure (indoor tobacco smoke, crowding, and cooking fuels, cooking place) among enrolled children. Where the acute asthma exacerbation will be suspected, physicians will assess the lung condition of the enrolled sick children using stethoscope and peak flow-meter. The lung function of children will be measured using spirometry, hyper-reactivity against common allergens will be performed using skin prick methods, exercise challenge test will be performed to understand the airway hyperresponsiveness, and blood eosinophil count determine the eosinophil level in the peripheral blood.

DETAILED DESCRIPTION:
Background: Respiratory syncytial virus (RSV) is the most common cause of childhood illness which attack the lower respiratory tract and develop bronchitis and pneumonia. Approximately 70% of infants are infected with RSV during their first year of life, and almost all children are infected at least once by 2 years of age (Wu & Hartert, 2011).

Each year, an estimated 33·1 million episodes of RSV-associated acute lower respiratory infections occur among under-five children globally, leading to 3·2 million hospitalizations and 118,200 deaths (Ting Shi & Acacio, 2017). The burden of RSV-associated severe acute lower respiratory tract infection is 10 times higher in developing countries compared to that in developed countries (36.1 per 1000 life birth vs 3.2 per 1000 life birth, respectively).

In addition to acute mortality and morbidity, RSV infection has a long-term effect on children's health (Jat & Kabra, 2017; Kneyber, Steyerberg, de Groot, & Moll, 2000). RSV infection can induce a state of bronchial hyper-reactivity that has an association with the development of asthma in later life (Balfour-Lynn, 1996), which, in turn, is a major risk factor of chronic obstructive pulmonary disease in adulthood (Svanes et al., 2010).. The prevalence of wheezing and asthma were reported two times higher in the children who had RSV bronchitis in infancy compared with children without a history of bronchiolitis during infancy (Sigurs et al., 2010). In a report, it was shown that among the children who experienced asthma by school age, 31% of them had healthcare visits in infancy due to respiratory diseases (Wu & Hartert, 2011). The severity of the RSV associated illness was reported as an additive factor for asthma risk. Hartert et, al., reported that asthma prevalence was two times higher in the infants who were hospitalized for RSV infection compared to the other who received care at the outdoor department (Wu & Hartert, 2011). In the mouse model, it was found that viral infection in neonatal rats delayed the growth of secondary septa, decreased the alveolar surface density by 14 to 26%, and reduced the diameter of terminal bronchioles by 11 and 20% (Castleman, Sorkness, Lemanske, Grasee, & Suyemoto, 1988). However, there is no data on the effect of RSV infection on the lung of neonates. In human, the lung remains premature at birth and continue to develop for 2-3 years postnatally and can be assumed that the impact of RSV infection during early infancy would be very severe.

Collecting clinical samples from young infants and lack of appropriate diagnostic to detect RSV virus are the major obstacles to study RSV infection in developing countries. No study from developing countries has investigated the long-term effect of RSV infections incurred during the young infant period. It is assumed that the long-term effect of RSV infection might be more intense if infection occurs during this period, as the lungs of newborns continue to develop for the first several months of life.

Recently, a study aimed to determine the etiology of young infant infection at five centers of three South Asian countries (Bangladesh, India, and Pakistan). This study identified 474 young infants who had laboratory-confirmed RSV infection; additionally, this study tested specimens from 1,873 age and sex-matched healthy infants, which were found to be negative for RSV. The current age of that cohort is between 5 and 7 years, which provides a unique opportunity to gather information on the long-term effect of RSV infection in a large number of laboratory-confirmed cases at a low cost.

Given the relative frequency and impact of RSV infection in developing healthcare settings, should the investigators identify a high prevalence of subsequent wheeze and asthma the potential benefit of interventions to reduce RSV will be enhanced. In addition, this study will have the following supplementary benefits (1) the ability to report the feasibility to identify wheeze frequency by self-reporting in South Asian populations, (2) the feasibility and outcomes of tests that are utilized to support the diagnosis of asthma and other respiratory diseases in children, i.e. skin prick tests, Eosinophil count and spirometry.

Research Questions: The overarching aim of this study is to understand the long-term effect on child health of RSV infection occurring in the first two months of life. Therefore, through this study, the investigators aim to investigate the following research questions:

1. Is there an association between RSV infection in the first two months of life and development of asthma later in childhood?
2. Is the lung function of children who had RSV infection in the first 2 months of life lower than that of children who did not have RSV infection?
3. Is there an association between RSV infection in the first two months of life and physical development in childhood?
4. Are risk factors for childhood asthma different for the children who had RSV infection in the first two months of life than others without RSV infection at the same age?

Methodologies: The investigators have identified sites of the Aetiology of Neonatal Sepsis in South Asia (ANISA) study, two in Pakistan and one each in Bangladesh and India to implement this study. Health workers will visit the households of eligible children. Children whose parents provide consent will be visited three times in one year period, at baseline, after six months and the end of the year. In the first visit, a member of the research team will explain the study objectives and procedures to one of the family members (primarily the mother) of the eligible children to provide consent for enrolling the children in the study, the parents of the enrolled children will be interviewed using a structured questionnaire to record the current and previous health status of children. Study team members will remain blind about the RSV infectious status of the children to avoid enrollment bias. To ascertain asthma and wheeze, parents will be inquired about breathing difficulties of the children using a questionnaire designed by the International Study of Allergies and Asthma in Childhood (ISAAC), dermatitis will be defined by the criteria provided by The U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis. It was previously reported that terms such as ''wheeze'' and ''difficulty in breathing'' used in the ISAAC questionnaire have little validity when comparing clinical cases between parents and also between clinicians, and the conceptual understandings of ''wheeze'' for parents of children with reported wheeze are different from definitions used in epidemiology (Bisgaard & Szefler, 2007). To reduce the differences in patient responses, the research team will provide a video demonstration of wheeze and asthma-like symptoms to the parents before introducing the questionnaire. They will also introduce a child "case card" to the parents and request to record the wheezing episodes of their enrolled children using this case card. Additionally, they will also request the parents to reach team (over the phone) if they notice wheezing sound to their children, a research team will visit the symptomatic children and perform a physical assessment of the child using auscultation and peak flowmetry. The research team will return to the families after six months to emphasize the use of the case card for recording wheeze episodes and also refer the children to the health facilities for physical assessment (spirometry, exercise challenge test, skin prick test, and eosinophil count test and anthropometric measurements). In the health facilities, physicians will perform afore mention tests and procedures. The research team will return to the families again after one year of the first visit and collect the "case card" from where they will record the number of wheeze/asthma episode occurred in the last one year (follow-up period).

ELIGIBILITY:
Inclusion Criteria:

RSV group

* Child was enrolled in the ANISA study
* Child had RSV infection in the first two months of life Non-RSV group
* Child was enrolled in the ANISA study
* Child provided respirator samples in the first two months of life
* Child was illness-free during the first two months of life
* RSV was not detected in the respiratory samples

Exclusion Criteria:

• Caregiver of the child is unwilling to participate in the study

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Between 2011 and 2015, ANISA study team members enrolled 56,987 newborns in four study sites. All the suspected sick infants were referred to the health facilities where study physicians assessed the infants using the criteria of possible serious bacterial. Infants who were identified as sick were advised to provide respiratory samples (oropharyngeal and nasopharyngeal swabs). Total 6,394 respiratory samples were collected from 5,350 ill infants, 433 infants were positive for RSV. Additionally, ANISA study team collected respiratory specimens from 1587 age and sex-matched healthy children who did not have any clinical sign of illness at the time of specimens collected and were also remain apparently healthy during both seven days prior to and seven days following sample collection. All these children are eligible to enroll in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Asthma among the children | at the age of 6-7 years of the enrolled children
  Caregiver reported three or more episodes of wheezing in the past 12 months OR One or more episode of wheeze and repeated cough during the night when the child did not have a cold or chest infection

SECONDARY OUTCOMES:
Maximum forced expiratory air volume in one second (FEV1) | at the age of 6-7 years of the children
  Lung function of the enrolled children will be measured using spirometry. Maximum forced expiratory air volume in one second will be reported
Hyperreactivity against allergens | at the age of 6-7 years of the children
  Skin prick test will be perform against common allergens to measure the hyperreactivity of the skin against those allergens
Height of the children | at the age of 6-7 years of the children
  Height of the children in meter
Weight of the children | at the age of 6-7 years of the children
  Weight of the children in Kilogram

IPD SHARING:
Plan to Share IPD: No
The personal information will be codified and the linkage data will not share with any other organization

REFERENCES:
- [Result] Balfour-Lynn IM. Why do viruses make infants wheeze? Arch Dis Child. 1996 Mar;74(3):251-9. doi: 10.1136/adc.74.3.251. No abstract available. PMID 8787436
- [Result] Bisgaard H, Szefler S. Prevalence of asthma-like symptoms in young children. Pediatr Pulmonol. 2007 Aug;42(8):723-8. doi: 10.1002/ppul.20644. PMID 17598172
- [Result] Castleman WL, Sorkness RL, Lemanske RF, Grasee G, Suyemoto MM. Neonatal viral bronchiolitis and pneumonia induces bronchiolar hypoplasia and alveolar dysplasia in rats. Lab Invest. 1988 Sep;59(3):387-96. PMID 3411939
- [Result] Jat KR, Kabra SK. Wheezing in children with viral infection & its long-term effects. Indian J Med Res. 2017 Feb;145(2):161-162. doi: 10.4103/ijmr.IJMR_1459_16. No abstract available. PMID 28639590
- [Result] Kneyber MCJ, Steyerberg EW, de Groot R, Moll HA. Long-term effects of respiratory syncytial virus (RSV) bronchiolitis in infants and young children: a quantitative review. Acta Paediatr. 2000 Jun;89(6):654-60. doi: 10.1080/080352500750043945. PMID 10914957
- [Result] Leung R, Ho P. Asthma, allergy, and atopy in three south-east Asian populations. Thorax. 1994 Dec;49(12):1205-10. doi: 10.1136/thx.49.12.1205. PMID 7878553
- [Result] Sigurs N, Aljassim F, Kjellman B, Robinson PD, Sigurbergsson F, Bjarnason R, Gustafsson PM. Asthma and allergy patterns over 18 years after severe RSV bronchiolitis in the first year of life. Thorax. 2010 Dec;65(12):1045-52. doi: 10.1136/thx.2009.121582. Epub 2010 Jun 27. PMID 20581410
- [Result] Siti Nadzrah Y, Zulkiflee AB, and Prepageran N. Common Aeroallergens by Skin Prick Test among the Population in Two Different Regions.Primary Healthcare 5: 206, 2015.
- [Result] Subbarao P, Mandhane PJ, Sears MR. Asthma: epidemiology, etiology and risk factors. CMAJ. 2009 Oct 27;181(9):E181-90. doi: 10.1503/cmaj.080612. Epub 2009 Sep 14. No abstract available. PMID 19752106
- [Result] Svanes C, Sunyer J, Plana E, Dharmage S, Heinrich J, Jarvis D, de Marco R, Norback D, Raherison C, Villani S, Wjst M, Svanes K, Anto JM. Early life origins of chronic obstructive pulmonary disease. Thorax. 2010 Jan;65(1):14-20. doi: 10.1136/thx.2008.112136. Epub 2009 Sep 2. PMID 19729360
- [Result] Shi T, McAllister DA, O'Brien KL, Simoes EAF, Madhi SA, Gessner BD, Polack FP, Balsells E, Acacio S, Aguayo C, Alassani I, Ali A, Antonio M, Awasthi S, Awori JO, Azziz-Baumgartner E, Baggett HC, Baillie VL, Balmaseda A, Barahona A, Basnet S, Bassat Q, Basualdo W, Bigogo G, Bont L, Breiman RF, Brooks WA, Broor S, Bruce N, Bruden D, Buchy P, Campbell S, Carosone-Link P, Chadha M, Chipeta J, Chou M, Clara W, Cohen C, de Cuellar E, Dang DA, Dash-Yandag B, Deloria-Knoll M, Dherani M, Eap T, Ebruke BE, Echavarria M, de Freitas Lazaro Emediato CC, Fasce RA, Feikin DR, Feng L, Gentile A, Gordon A, Goswami D, Goyet S, Groome M, Halasa N, Hirve S, Homaira N, Howie SRC, Jara J, Jroundi I, Kartasasmita CB, Khuri-Bulos N, Kotloff KL, Krishnan A, Libster R, Lopez O, Lucero MG, Lucion F, Lupisan SP, Marcone DN, McCracken JP, Mejia M, Moisi JC, Montgomery JM, Moore DP, Moraleda C, Moyes J, Munywoki P, Mutyara K, Nicol MP, Nokes DJ, Nymadawa P, da Costa Oliveira MT, Oshitani H, Pandey N, Paranhos-Baccala G, Phillips LN, Picot VS, Rahman M, Rakoto-Andrianarivelo M, Rasmussen ZA, Rath BA, Robinson A, Romero C, Russomando G, Salimi V, Sawatwong P, Scheltema N, Schweiger B, Scott JAG, Seidenberg P, Shen K, Singleton R, Sotomayor V, Strand TA, Sutanto A, Sylla M, Tapia MD, Thamthitiwat S, Thomas ED, Tokarz R, Turner C, Venter M, Waicharoen S, Wang J, Watthanaworawit W, Yoshida LM, Yu H, Zar HJ, Campbell H, Nair H; RSV Global Epidemiology Network. Global, regional, and national disease burden estimates of acute lower respiratory infections due to respiratory syncytial virus in young children in 2015: a systematic review and modelling study. Lancet. 2017 Sep 2;390(10098):946-958. doi: 10.1016/S0140-6736(17)30938-8. Epub 2017 Jul 7. PMID 28689664
- [Result] Wu P, Hartert TV. Evidence for a causal relationship between respiratory syncytial virus infection and asthma. Expert Rev Anti Infect Ther. 2011 Sep;9(9):731-45. doi: 10.1586/eri.11.92. PMID 21905783